CLINICAL TRIAL: NCT00067301
Title: PUFA Augmentation in Treatment of Major Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21AT001077 (NIH); GertsikL
Record Dates: First submitted 2003-08-14; First posted 2003-08-15 (Estimated); Last update posted 2008-01-25 (Estimated); Status verified 2008-01

CONDITIONS: Major Depression
Keywords: depression; citalopram; Celexa; Polyunsaturated Fatty Acids; omega-3; EPA; antidepressants
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Fatty Acids, Unsaturated; Citalopram

INTERVENTIONS:
Drug: Polyunsaturated Fatty Acids (PUFA)
Drug: Citalopram

SUMMARY:
The purpose of this study is to determine if omega-3 fatty acid EPA will enhance and speed up response to antidepressant therapy with Celexa (Citalopram) in people suffering from Major Depressive Disorder. All patients will receive Celexa, 50% will receive EPA, 50% placebo EPA.

DETAILED DESCRIPTION:
As per brief summary

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-IV criteria for current major depression, and have a HAM-D (21 item) score of > 17
* Male or female who, if of child-bearing potential, agrees to use effective contraception including the regular use of contraceptive pills, intra-uterine devices, barrier methods or abstinence
* Age between 18 and 65
* Capable of giving informed consent

Exclusion Criteria:

* Diagnosis of schizophrenia, schizophreniform disorder, schizoaffective disorder, schizotypal disorder, psychotic depression or bipolar disorders
* Current drug or alcohol abuse or dependence, or history of drug or alcohol abuse or dependence within the previous 6 months
* Unstable medical or neurological conditions that are likely to interfere with the treatment of depression
* History of allergy to citalopram or ProEPA, finfish or shellfish
* History of failure of response to citalopram, as documented by an adequate trial of the medication [defined as having been treated with the medication at a dose level typically regarded as adequate (i.e., 40 mg of citalopram per day) for at least 6 weeks]
* History of seizure disorder
* Pregnancy
* Currently on psychotropic medications including antidepressants or neuroleptics
* Active suicidal ideation or other safety issues determined by the clinician to not be suitable for inclusion in the study
* Exposure to treatment with fluoxetine or MAOIs in the previous two months
* Patients on anticoagulant therapy
* Patients with a dietary intake of > 3.0g total omega-3 PUFA/day at baseline

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-09; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lev Gertsik, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center Dept. of Psychiatry, Los Angeles, California, United States

REFERENCES:
- [Derived] Appleton KM, Voyias PD, Sallis HM, Dawson S, Ness AR, Churchill R, Perry R. Omega-3 fatty acids for depression in adults. Cochrane Database Syst Rev. 2021 Nov 24;11(11):CD004692. doi: 10.1002/14651858.CD004692.pub5. PMID 34817851